CLINICAL TRIAL: NCT00190762
Title: A Randomized Phase 3 Trial Comparing ALIMTA Plus Best Supportive Care Versus Best Supportive Care Alone in Previously Treated Patients With Locally Advanced or Metastatic Malignant Pleural Mesothelioma
Brief Title: A Study Comparing Pemetrexed Plus Best Supportive Care Versus Best Supportive Care Alone in the Treatment of Mesothelioma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5362; H3E-MC-JMEW
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Mesothelioma
MeSH Terms: conditions — Mesothelioma | interventions — Pemetrexed

INTERVENTIONS:
Drug: Pemetrexed

SUMMARY:
Based on results from earlier clinical trials, Pemetrexed may have antitumor activity as a first-line agent in the treatment of mesothelioma. Given this, it is hypothesized that Pemetrexed may be active in second-line mesothelioma in which the standard treatment is best supportive care. This study will compare survival of previously treated patients with malignant pleural mesothelioma who receive Pemetrexed plus best supportive care to the survival of similar patients who receive best supportive care alone.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of mesothelioma of the pleura.
* received only one prior systemic chemotherapy regimen for advanced or metastatic disease
* Performance status of 70 or higher on the Karnofsky Performance Status Scale
* Males or females at least 18 years of age
* Adequate organ function

Exclusion Criteria:

* Active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy
* Pregnancy or breastfeeding
* Brain metastasis
* Prior treatment with Pemetrexed
* Inability or unwillingness to take folic acid or vitamin B12 supplementation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 2001-10; Study Completion 2005-11

PRIMARY OUTCOMES:
The primary objective of this study is to compare the overall survival following treatment with Pemetrexed plus best supportive care versus best supportive care alone

SECONDARY OUTCOMES:
To characterize and compare the toxicities of Pemetrexed/best supportive care and best supportive care alone in this patient population;to determine the objective-tumor response rate
to compare time to event efficacy variables of both arms including:duration of response,time to objective tumor response,time to treatment failure,time to documented disease progression,progression-free survival
to compare changes in the average symptom burden index between the Pemetrexed/best supportive care and best supportive care arms

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Monday-Friday 9am-5pm Eastern time (UTC/GMT-5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9:00 AM - 5:00 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician, Ottawa, Ontario, Canada